CLINICAL TRIAL: NCT05683925
Title: Effect of Transcutaneous Auricular Vagus Nerve Stimulation at 25Hz and 100Hz on Levodopa Responsive and Non-responsive Gait Characteristics in Parkinson's Disease- a Motion Sensor Study
Brief Title: Effect of Transcutaneous Auricular Vagus Nerve Stimulation on Gait Characteristics in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Maja Kojović, assoc. prof., University Medical Centre Ljubljana
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 012052/2020/2
Record Dates: First submitted 2022-12-19; First posted 2023-01-13 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic
Keywords: parkinson's disease; taVNS; motion sensors
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Participants and study overview In this randomised placebo controlled trial, the investigators will include 30 PD patients with HY>2 and L-dopa unresponsive gait characteristics. Each participant will complete 1 visit, during which the instrumented stand and walk test will be repeated 16 times. The baseline measurement will be followed by three different stimulation conditions sham VNS (sVNS), taVNS at 25Hz (taVNS25) and taVNS a 100Hz (taVNS100). sVNS, taVNS25 and taVNS100 in a randomized order. To enhance gait disturbances, the participants will preform iSAW during each condition twice in silence and twice while simultaneously performing calculations around.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Noninvasive electrostimulation will be applied to the left ear. taVNS will be applied to the cyma conchae and sVNS will be applied to the earlobe - participants will not be told which is the active and which is the sham condition. Both taVNS and sVNS were applied through the Nemos® electrode. The intensity for each separate stimulation will be adjusted for each participant at the beginning of the experiment. For each condition, the electrode will be placed in the ear by a third person and the ear will be covered by cotton pads and an EEG cap to hide the electrode position from the experimenter. The order of stimulation will not be revealed until the automated data and statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- baseline (No Intervention): Participants will receive no stimulation, the electrode will be placed in the ear in a random position and turned off. Participants will complete 4 instrumented stand and walk tests - 2 without performing calculations and 2 with performing calculations aloud.
- taVNS100 (Active Comparator): Noninvasive electrostimulation will be applied to the left cyma conchae through the Nemos® electrode at 100Hz. Participants will complete 4 instrumented stand and walk tests - 2 without performing calculations and 2 with performing calculations aloud.
  Interventions: Device: Noninvasive transcutaneous auricular vagus nerve stimulation at 100Hz
- taVNS25 (Active Comparator): Noninvasive electrostimulation will be applied to the left cyma conchae through the Nemos® electrode at 25Hz. Participants will complete 4 instrumented stand and walk tests - 2 without performing calculations and 2 with performing calculations aloud.
  Interventions: Device: Noninvasive transcutaneous auricular vagus nerve stimulation at 25Hz
- sVNS (Sham Comparator): Noninvasive electrostimulation will be applied to the left earlobe through the Nemos® electrode at 25Hz. Participants will complete 4 instrumented stand and walk tests - 2 without performing calculations and 2 with performing calculations aloud.
  Interventions: Device: Noninvasive transcutaneous earlobe stimulation at 25Hz

INTERVENTIONS:
Device: Noninvasive transcutaneous auricular vagus nerve stimulation at 100Hz — Noninvasive electrostimulation will be applied to the left cyma conchae through the Nemos® electrode with the following parameters: square-shaped pseudobiphasic pulse, interpulse duration 80μs, pulse width 300μs, pulse intensity 0,1mA above the perceptual threshold at 100Hz. The intensity for each separate stimulation will be adjusted for each participant at the beginning of the experiment.
  Other Names: taVNS100
  Arms: taVNS100
Device: Noninvasive transcutaneous auricular vagus nerve stimulation at 25Hz — Noninvasive electrostimulation will be applied to the left cyma conchae through the Nemos® electrode with the following parameters: square-shaped pseudobiphasic pulse, interpulse duration 80μs, pulse width 300μs, pulse intensity 0,1mA above the perceptual threshold at 25Hz. The intensity for each separate stimulation will be adjusted for each participant at the beginning of the experiment.
  Other Names: taVNS25
  Arms: taVNS25
Device: Noninvasive transcutaneous earlobe stimulation at 25Hz — Noninvasive electrostimulation will be applied to the left earlobe through the Nemos® electrode with the following parameters: square-shaped pseudobiphasic pulse, interpulse duration 80μs, pulse width 300μs, pulse intensity 0,1mA above the perceptual threshold at 25Hz. The intensity for each separate stimulation will be adjusted for each participant at the beginning of the experiment.
  Other Names: sVNS
  Arms: sVNS

SUMMARY:
In this randomised placebo-controlled trial, the investigators will include 30 PD (Parkinson's disease) patients with HY (Hoehn Yahr stage) >2 and L-dopa unresponsive gait characteristics. Each participant will receive taVNS at 25Hz, taVNS at 100Hz and sham VNS (sVNS). During each stimulation, different gait characteristics will be measured with wearable insertion motion sensors.

DETAILED DESCRIPTION:
Participants and study overview:

In this randomised placebo-controlled trial, the investigators will include 30 PD patients with HY>2 and L-dopa unresponsive gait characteristics. Each participant will complete 1 visit, during which the instrumented stand and walk test will be repeated 16 times. The baseline measurement will be followed by three different stimulation conditions sham VNS (sVNS), taVNS at 25Hz (taVNS25) and taVNS a 100Hz (taVNS100). sVNS, taVNS25 and taVNS100 in a randomized order. To enhance gait disturbances, the participants will perform iSAW during each condition twice in silence and twice while simultaneously performing calculations around.

Instrumented stand and walk test (iSAW):

To perform iSAW, participants will first stand still for 30s, after which they will start walking in a straight line for 7m, turn and walk back to the start. The participants will be equipped with 6 inertion Opal ® motion sensors (on both feet, both wrists, on the lumbar back and on their sternum). For the laud counting iSAW condition (iSAW-C), the participants will perform iSAW as described above while also counting backwards by 3 from numbers above 100.

TaVNS:

Noninvasive electrostimulation will be applied to the left ear. taVNS will be applied to the cyma conchae and sVNS will be applied to the earlobe. Both taVNS and sVNS were applied through the Nemos® electrode with the following parameters: square-shaped pseudobiphasic pulse, interpulse duration 80μs, pulse width 300μs, pulse intensity 0,1mA above the perceptual threshold (figure 1). taVNS25 and sVNS will be applied at 25Hz and taVNS100 will be applied at 100Hz. The intensity for each separate stimulation will be adjusted for each participant at the beginning of the experiment. For each condition, the electrode will be placed in the ear by a third person and the ear will be covered by cotton pads and an EEG cap to hide the electrode position from the experimenter. The order of stimulation will not be revealed until the automated data and statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* HYstage >2
* L-dopa unresponsive gait characteristics present, preferably with history of freezings

Exclusion Criteria:

* unable to walk for 50m
* unable to follow simple commands due to hearing loss/cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Arm Swing Velocity | This will be measured acutely, e. i. during taVNS/sVNS and compared to baseline measurements.
  The average velocity of upper extremities in degrees per second as produced by the Mobility Lab software.
Arm Range of Motion | This will be measured acutely, e. i. during taVNS/sVNS and compared to baseline measurements.
  The average wrist range of motion in degrees as produced by the Mobility Lab software.
Stride Length | This will be measured acutely, e. i. during taVNS/sVNS and compared to baseline measurements.
  The average stride length in m as produced by the Mobility Lab software.
Gait Speed | This will be measured acutely, e. i. during taVNS/sVNS and compared to baseline measurements.
  The average speed of gait in m/s as produced by the Mobility Lab software.
Arm Range of Motion Asymmetry | This will be measured acutely, e. i. during taVNS/sVNS and compared to baseline measurements.
  The average difference between left and right arm range of motion in degrees as produced by the Mobility Lab software.
Anticipatory Postural Adjustment (APA) duration | This will be measured acutely, e. i. during taVNS/sVNS and compared to baseline measurements.
  The average duration of anticipatory postural adjustments in seconds as produced by the Mobility Lab software.
APA First step Duration | This will be measured acutely, e. i. during taVNS/sVNS and compared to baseline measurements.
  The average duration of the first detected step in seconds as produced by the Mobility Lab software.
APA First Step range of motion | This will be measured acutely, e. i. during taVNS/sVNS and compared to baseline measurements.
  The average range of motion of the first detected step as produced by the Mobility Lab software.

CONTACTS AND LOCATIONS:
Overall Officials: Maja Kojović, MD, PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- Neurology Department, UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share the anonymised data with researchers upon request.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Upon request after study publication.
Access Criteria: Data will be shared with researchers upon reasonable request.